CLINICAL TRIAL: NCT07403825
Title: Efficacy of Faricimab in Patients With Subretinal Hyperreflective Material Associated With Type 2 or Mixed Neovascular Membranes Assessed by Multimodal Imaging
Brief Title: Efficacy of Faricimab in Patients With Subretinal Hyper-reflective Material
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Biobizkaia Health Research Institute (Other Government)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FARIDUO
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Macular Degeneration, Age Related
MeSH Terms: conditions — Macular Degeneration | interventions — Injections; faricimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vabysmo (Experimental): Experimental arm
  Interventions: Drug: Vabysmo 6 MG in 0.05 ML Injection

INTERVENTIONS:
Drug: Vabysmo 6 MG in 0.05 ML Injection — The study drug, Faricimab (Vabysmo®), will be administered at a dose of 6 mg/0.05 ml, by intravitreal injection, following the indications in the product's technical data sheet.
  Other Names: Faricimab

SUMMARY:
Whose aim is to:

Determine the percentage of patients with resolution of subretinal hyperreflective material (SHRM) at week 16.

This study is intended to be performed in the ophthalmology departments or ophthalmology clinics of the participating sites, located in Spain.

Macular degeneration is an eye disease characterised by progressive damage to the macula leading to a loss of central vision. There are two types of macular degeneration, dry and wet or exudative. The prevalence of the latter in Spain is 1.9% in people aged 65 and over. Among the subtypes of macular neovascularisation (MNV), type 2 is rare (9%), with the majority being mixed type 1 and 2 cases (13.5%). SHRM is present in about 77% of eyes with neovascular age-related macular degeneration (AMD).

Different anti-VEGF (vascular endothelial growth factor) drugs have been used for the treatment of type 2 and mixed 1 and 2 types of MNV. Following treatment, a reduction in SHRM has been observed, although results between studies vary between 34% and 56%. Improvements in best-corrected visual acuity are also achieved in eyes with type 2 MNV with anti-VEGF therapy.

DETAILED DESCRIPTION:
In this phase IV, multicentre, prospective, longitudinal, uncontrolled, prospective clinical trial, patients will be administered the marketed drug Vabysmo®, whose active ingredient is Faricimab. It is an injectable humanised antibody that acts on two different pathways, by neutralising both Ang-2 and VEGF-A. It is indicated for the treatment of adult patients with neovascular AMD, patients with visual impairment due to diabetic macular oedema or patients with visual impairment due to macular oedema secondary to retinal vein occlusion. It may also have a role in stabilising neovascular membranes, as well as a possible antifibrotic effect, reducing the presence of SHRM, after seeing real clinical cases with subretinal haemorrhage and very good response to this drug, probably due to its dual inhibition with Ang-2 suppression.

ELIGIBILITY:
Inclusion Criteria:

* People aged 50 and over.
* Diagnosed with bilateral or unilateral AMD.
* Eyes with SHRM and type 2 or mixed (type 1 and 2) neovascular membrane.
* Näive eyes treated with Faricimab following SmPC (summary of product characteristic).
* They agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Eyes with type 1, aneurysmal type 1 and type 3 MNV.
* Eyes with type 2 MNV and other macular diseases (myopia, posterior uveitis, systemic diseases, such as pseudoxanthoma elasticum).
* Eyes with ocular media opacity.
* Patients with other retinal diseases, such as central serous chorioretinopathy, diabetic retinopathy, retinal vascular occlusion, uveitis, myopic maculopathy or any other retinal disease that could compromise the best-corrected visual acuity and interfere with retinal parameters.
* Any neurological condition (including cognitive impairment, stroke, dementia, Parkinson, anxiety or schizophrenia) that, in the opinion of the investigator, would pose a risk to patient's safety or interfere with the assessment, procedures, or completion of the study.
* People who are participating or will participate in any type of clinical trial.
* Pregnant women.
* Breastfeeding women.
* Women* of childbearing potential who are unable or unwilling to use highly effective methods of contraception (bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices) from the start to the end of the study.

  * Woman of childbearing potential: considered as such if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), or has not undergone surgical sterilization (removal of ovaries and/or uterus).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
to assess the resolution of SHRM at week 16 | finish to the clinical trial
  The percentage of patients with resolution of SHRM at week 16.